CLINICAL TRIAL: NCT01913353
Title: A Randomized, Open-label Phase III Non-inferiority Trial to Compare Indicators of Efficacy for MVA-BN® Smallpox Vaccine to ACAM2000® in 18-42 Year Old Healthy Vaccinia-naïve Subjects
Brief Title: A Non-inferiority Trial to Compare MVA-BN® Smallpox Vaccine to ACAM2000®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: POX-MVA-006
Record Dates: First submitted 2013-07-26; First posted 2013-08-01 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: 18-42 Year Old Healthy Vaccinia-naïve Subjects
MeSH Terms: interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic; ACAM2000

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Two vaccinations; MVA BN ®; administered 4 weeks apart (Day 0 and Day 28) followed by a single vaccination of ACAM2000® vaccine 4 weeks after the second MVA BN® vaccination (Day 56).
  Interventions: Biological: MVA BN®; Biological: ACAM2000®
- Group 2 (Active Comparator): A single vaccination of ACAM2000® will be administered at Day 0.
  Interventions: Biological: ACAM2000®

INTERVENTIONS:
Biological: MVA BN® — 0.5 ml MVA BN® with a nominal titer of 1x10E8 TCID50, administered as a subcutaneous injection
  Other Names: IMVAMUNE; IMVANEX
  Arms: Group 1
Biological: ACAM2000® — 0.0025 ml ACAM2000®, consisting of 2.5-12.5x10E5 plaque forming units of live vaccinia virus (VACV). Picked up with a bifurcated needle and administered by the percutaneous route (scarification) using 15 jabs of that bifurcated needle.

SUMMARY:
To demonstrate the efficacy of MVA-BN® in terms of vaccinia-specific Plaque Reduction Neutralization Test (PRNT) antibody response and by showing that vaccination prior to administration of ACAM2000® results in an attenuated take.

DETAILED DESCRIPTION:
To demonstrate the efficacy of MVA-BN® by assessing non-inferiority of MVA-BN® compared to ACAM2000® in terms of vaccinia-specific Plaque Reduction Neutralization Test (PRNT) antibody response at the Peak Visits (Day 42 for Group 1 and Day 28 for Group 2) and by showing that vaccination with MVA-BN® prior to administration of ACAM2000® results in an attenuation of take.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, 18-42 years of age
2. The subject has read, signed and dated the Informed Consent, having been advised of the risks and benefits of the trial in a language understood by the subject and prior to performance of any trial specific procedure
3. Acceptable medical history by screening evaluation and physical examination
4. BMI greater or eaqual than 18.5 and smaller than 35
5. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at Screening and a negative urine or serum pregnancy test within 24 hours prior to each vaccination
6. WOCBP must have used an acceptable method of contraception for 28 days prior to the first vaccination, must agree to use an acceptable method of contraception during the trial, and must avoid becoming pregnant for at least 28 days after the last vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products)
7. Human Immunodeficiency Virus (HIV) antibody negative, hepatitis B surface antigen negative and negative antibody test to hepatitis C virus
8. White blood cells greater or eaqual than 2500/mm3 and smaller than 11,000/mm3
9. Hemoglobin within normal limits
10. Platelets greater or eaqual than lower normal limits
11. Adequate renal function defined as a calculated Creatinine Clearance (CrCl) greater than 60 ml/min as estimated by the Cockcroft-Gault equation
12. Adequate hepatic function in the absence of other evidence of significant liver disease defined as:

    * Total bilirubin greater than 1.5 x Upper Limit Normal (ULN)
    * Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) greater than 1.5 x ULN
    * Alkaline Phosphatase (Alk Phos) greater than 1.5 x ULN
13. Troponin I smaller than 2 x ULN
14. Electrocardiogram (ECG) without clinically significant findings, e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, atrioventricular node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions in a row, ST elevation consistent with ischemia

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Typical vaccinia scar
3. Known or suspected history of smallpox vaccination defined as visible vaccination scar or documentation of smallpox vaccination or as reported by the subject
4. History of vaccination with any poxvirus-based vaccine
5. History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject
6. History of or active immunodeficiency or immunosuppression caused by acquired or congenital diseases or caused by ongoing treatments such as chronic (greater than 14 days) high-dose corticosteroids (smaller than 5 mg prednisone [or equivalent] per day applied systemically, i.e. parenterally or orally), chronic or planned treatment with steroid eye drops or ointment at time of enrollment or radiation, or immunosuppressive drugs; low-dose corticosteroid topical products and nasal sprays used sporadically, i.e. pro re nata (according to circumstances) are permissible
7. Having had radiation or X-ray treatment (not routine X-rays) within the last 3 months
8. Post organ and bone-marrow transplant subjects whether or not receiving chronic immunosuppressive therapy
9. Eye surgery within 4 weeks prior to trial vaccination
10. History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid hormone replacement are not excluded
11. Uncontrolled serious infection, i.e. not responding to antimicrobial therapy
12. History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous site of cancer
13. History of keloid formation
14. History or clinical manifestation of severe hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders
15. History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor
16. Chest pain (that is diagnosed as cardiac related) or trouble breathing on exertion
17. Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's Risk Assessment Tool: http://hin.nhlbi.nih.gov/atpiii/calculator.asp NOTE: This criterion applies only to subjects 20 years of age and older
18. History of an immediate family member (father, mother, brother, or sister) who has had onset of ischemic heart disease before the age of 50 years
19. Clinically significant psychological disorder not adequately controlled by medical treatment
20. Active or history of chronic alcohol abuse and/or intravenous and/or nasal drug abuse (within the past 6 months)
21. History of anaphylaxis or any severe allergic reaction or serious adverse reaction to a vaccine
22. Eczema of any degree or history of eczema
23. People with active atopic dermatitis (AD) [characterized by pruritus, eczematous lesions, xerosis (dry skin), and lichenification (thickening of the skin and an increase in skin markings] or with a history of AD
24. People with chronic exfoliative skin disorders/conditions
25. People with active current Varicella zoster, Herpes zoster, impetigo, uncontrolled acne, Darier's disease or any acute skin disorders of large magnitude, e.g., laceration requiring sutures
26. People with a tattoo that covers the vaccination injection area (preventing assessment of the area and interfering with a vaccination site photograph)
27. Having received any vaccinations or planned vaccinations with a live vaccine within 28 days prior to or after trial vaccination
28. Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior to or after trial vaccination
29. Administration or planned administration of immunoglobulins and/or any blood products during a period starting from three months prior to administration of the vaccine and ending at trial conclusion
30. Use of any investigational or non-registered drug or vaccine other than the trial vaccines within 28 days preceding the first dose of the trial vaccine or planned administration of such a drug /vaccine during the trial period
31. Blood donation for the duration of the trial
32. Acute disease (illness with or without a fever) at the time of enrollment
33. Temperature ≥ 100.4°F (38.0°C) at the time of enrollment
34. Known household contacts with, or occupational exposure (other than minimal contact) to any of the following:

    * Pregnant women
    * Children <12 months of age
    * People with eczema or a history of eczema
    * People with active AD or history of AD
    * People with chronic exfoliative skin disorders/conditions
    * People with active Varicella zoster, Herpes zoster, impetigo, uncontrolled acne, Darier's disease or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn with areas greater than 2×2 cm
    * People with active or recent immunodeficiency disease or use of immunosuppressive medications, for example: have or take medication for HIV, AIDS, leukemia, lymphoma, or chronic liver problem, have or take medication for Crohn's disease, lupus, arthritis, or other immune disease; have had radiation or X-ray treatment (not routine X-rays) within the last 3 months; have ever had a bone-marrow or organ transplant (or take medication for that ); or have another problem that requires steroids, prednisone or a cancer drug for treatment
    * People having had eye surgery within the last 4 weeks
35. Known allergy to MVA-BN® vaccine or any of its constituents, e.g. tris(hydroxymethyl)-amino methane, including known allergy to egg or aminoglycoside (gentamycin)
36. Known allergies to ACAM2000® and its diluents including polymyxin B sulfate, neomycin sulfate, and phenol
37. Known allergies to vaccinia immunoglobulin (VIG) including thimerosal or previous allergic reaction to immunoglobulins
38. Known allergies to cidofovir, sulfa drugs, or probenecid
39. Trial personnel

Ages: 18 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 440 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip R Pittman, MD, MPH, Principal Investigator — US Army Medical Research Institute of Infectious Diseases
Locations (1):
- Brian Allgood Army Community Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Pittman PR, Hahn M, Lee HS, Koca C, Samy N, Schmidt D, Hornung J, Weidenthaler H, Heery CR, Meyer TPH, Silbernagl G, Maclennan J, Chaplin P. Phase 3 Efficacy Trial of Modified Vaccinia Ankara as a Vaccine against Smallpox. N Engl J Med. 2019 Nov 14;381(20):1897-1908. doi: 10.1056/NEJMoa1817307. PMID 31722150

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started (Randomized including subjects not vaccinated) | 221 | 219
Completed (Active trial phase) | 189 | 204
Not Completed | 32 | 15
Not completed — Adverse Event | 2 | 0
Not completed — Physician Decision | 0 | 2
Not completed — Withdrawal by Subject | 20 | 6
Not completed — multiple reasons | 10 | 7

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Group 1: Two vaccinations; MVA BN ®; administered 4 weeks apart (Day 0 and Day 28) followed by a single vaccination of ACAM2000® vaccine 4 weeks after the second MVA BN® vaccination (Day 56).
  MVA BN®: 0.5 ml MVA BN® with a nominal titre of 1x10E8 TCID50, administered as a subcutaneous injection
  ACAM2000®: 0.0025 ml ACAM2000®, consisting of 2.5-12.5x10E5 plaque forming units of live vaccinia virus (VACV). Picked up with a bifurcated needle and administered by the percutaneous route (scarification) using 15 jabs of that bifurcated needle.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 220 | 213 | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.5 (4.77) | 23.4 (4.58) | 23.5 (4.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 29 | 68
  Male | 181 | 184 | 365
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 40 | 94
  Not Hispanic or Latino | 166 | 173 | 339
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 6 | 14
  Asian | 14 | 12 | 26
  Native Hawaiian or Other Pacific Islander | 5 | 3 | 8
  Black or African American | 48 | 40 | 88
  White | 126 | 136 | 262
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 16 | 35
Region of Enrollment [Number; unit: participants]
  South Korea | 220 | 213 | 433

OUTCOME MEASURES:

1. Primary Outcome: Plaque Reduction Neutralization Test (PRNT) Geometric Mean Titer (GMT) at the Peak Visits
Description: GMT based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of 1.
Time Frame: Day 42 for Group 1 and Day 28 for Group 2
Population: Per-protocol Set for Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- Group 1: Two vaccinations; MVA-BN ®; administered 4 weeks apart (Day 0 and Day 28) followed by a single vaccination of ACAM2000® vaccine 4 weeks after the second MVA-BN® vaccination (Day 56).
  MVA-BN®: 0.5 ml MVA-BN® with a nominal titer of 1x10E8 TCID50, administered as a subcutaneous injection
  ACAM2000®: 0.0025 ml ACAM2000®, consisting of 2.5-12.5x10E5 plaque forming units of live vaccinia virus (VACV). Picked up with a bifurcated needle and administered by the percutaneous route (scarification) using 15 jabs of that bifurcated needle.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
Titer | 153.5 [134.3 to 175.6] | 79.3 [67.1 to 93.8]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Non-Inferiority — The non-inferiority margin to show that Group 1 (after 2 doses of MVA-BN) is non-inferior to Group 2 (after 1 dose of ACAM2000) in terms of PRNT GMTs at the respective peak visit (Week 6 in Group 1 / Week 4 in Group 2) was predefined as '1/2 (i.e. 0.5)' for the GMT ratio (Group 1 / Group 2); GMT Ratio (Group 1 / Group 2) = 1.935, 95% CI 2-sided [1.562 to 2.397]

2. Primary Outcome: Maximum Lesion Area (MLA) in mm2 After Scarification With ACAM2000®
Description: The MLA was defined as the maximum of two measurements: the lesion area measured on Day 6-8 (after scarification) or the lesion area measured on Day 13-15 (after scarification). This was measured using the SilhouetteConnect camera system, and confirmed by the Independent Take Review Committee (ITRC).
Time Frame: Day 6-8, 13-15 after 3rd Vaccination for Group 1 and Day 6-8, 13-15 after 1st vaccination for Group 2
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm2 | 0.0 [0.0 to 2.0] | 76.0 [70.0 to 87.0]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority — Predefined threshold of clinical relevance for the area attenuation ratio (AAR): 40%; Area attenuation ratio (AAR) = 97.9, 95% CI 2-sided [96.6 to 98.3] — The AAR, i.e. the reduction in MLA [1 - MLA ratio (Group 1/Group 2)] after scarification was to be significantly above 40%. The MLA ratio and the corresponding 95% CI were based on the Hodges-Lehmann estimate of the shift for log-transformed MLAs

3. Secondary Outcome: Investigator-measured Maximum Lesion Diameter (MLD) in mm After Scarification With ACAM2000
Description: The MLD was defined as the largest major diameter measured across the lesion on Day 6-8 (after scarification) or Day 13-15 (after scarification)
Time Frame: Day 6-8 and Day 13-15 after ACAM2000 scarification
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm | 0.0 [0.0 to 2.0] | 11.0 [10.0 to 11.0]

4. Secondary Outcome: Investigator-measured Lesion Diameter in mm at Day 6-8 After Scarification With ACAM2000
Description: The lesion diameter at Day 6-8 was defined as the major lesion diameter measured on Day 6-8 (after scarification)
Time Frame: Day 6-8 after ACAM2000 scarification
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm | 0.0 [0.0 to 2.0] | 8.0 [8.0 to 9.0]

5. Secondary Outcome: Investigator-measured Lesion Diameter in mm at Day 13-15 After Scarification With ACAM2000
Description: The lesion diameter at Day 13-15 was defined as the major lesion diameter measured on Day 13-15 (after scarification)
Time Frame: Day 13-15 after ACAM2000 scarification
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm | 0.0 [0.0 to 0.0] | 10.0 [10.0 to 11.0]

6. Secondary Outcome: Individual Take as Classified by a Blinded Independent Take Review Committee (ITRC)
Description: Take was assessed as either full, partial, or absent take by the ITRC based on Day 6-8 evaluations following ACAM2000 vaccination using subject profiles that contained supportive data up to Day 14 following ACAM2000 vaccination (in accordance with the ITRC Charter).
Time Frame: Day 6-8 visit following ACAM2000 vaccination
Population: Per-protocol Set
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
percentage of subjects
  Full Take | 23.0 [16.8 to 30.2] | 92.5 [87.3 to 96.1]
  Partial Take | 23.0 [16.8 to 30.2] | 4.3 [1.8 to 8.8]
  Absent Take | 53.9 [46.0 to 61.7] | 1.9 [0.4 to 5.3]
  Missing | 0 [0.0 to 2.2] | 1.2 [0.2 to 4.4]

7. Secondary Outcome: Lesion Area in mm2 at Day 6-8 After Scarification With ACAM2000
Description: Lesion area was measured by the Investigator using the SilhouetteConnect camera system and confirmed by the blinded ITRC.
Time Frame: Day 6-8 after ACAM2000 scarification
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm2 | 0.0 [0.0 to 1.0] | 37.0 [33.0 to 42.0]

8. Secondary Outcome: Lesion Area in mm2 at Day 13-15 After Scarification With ACAM2000
Description: as for outcome 7
Time Frame: Day 13-15 after ACAM2000 scarification
Population: Per-protocol Set
Measure: Median (95% Confidence Interval); unit: mm2
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 165 | 161
mm2 | 0.0 [0.0 to 0.0] | 75.0 [69.0 to 85.0]

9. Secondary Outcome: Relationship to Vaccine of Any Serious Adverse Event (SAE)
Description: Presentation of SAEs by relationship to study vaccine
Time Frame: Within 38 weeks for Group 1 and 30 weeks for Group 2
Population: Full Analysis Set
Measure: Number; unit: Events
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 220 | 213
Events
  Unrelated/None | 4 | 2
  Unlikely | 1 | 1
  Possible | 0 | 0
  Probable | 0 | 0
  Definite | 0 | 0

10. Secondary Outcome: Intensity of Any Serious Adverse Event (SAE)
Description: Presentation of SAEs by intensity
Time Frame: Within 38 weeks for Group 1 and 30 weeks for Group 2
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 220 | 213
participants
  Mild: routine daily activity not impaired | 0 | 0
  Moderate: routine daily activity impaired | 0 | 0
  Severe: prevents routine daily activities | 1 | 1
  Life threatening | 4 | 2

11. Secondary Outcome: Incidence of Any Cardiac Sign or Symptom Indicating a Case of Myo-/Pericarditis, i.e. Adverse Events of Special Interest (AESIs)
Description: In this clinical trial, an AESI was defined as any cardiac sign or symptom developed since the first vaccination, any ECG changes determined to be clinically significant, or any cardiac enzyme results of Troponin I ≥ 2 x ULN.
Time Frame: Within 38 weeks for Group 1 and 30 weeks for Group 2
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Group 1, Period 1: after 1st dose of MVA-BN
- Group 1, Period 2: after second dose of MVA-BN
- Group 1, Period 3: after ACAM2000
- Group 2: ACAM2000
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 220 | 208 | 196 | 213
Participants | 2 | 2 | 3 | 4

12. Secondary Outcome: Related Grade >=3 Adverse Events
Description: Incidence of any Grade 3 or 4 adverse events (AEs) possibly, probably, or definitely related to the vaccine. Pooled solicited (general only) and unsolicited AEs.
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- Group 1, Period 2: after 2nd dose of MVA-BN
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 220 | 208 | 196 | 213
Participants | 3 | 2 | 3 | 22

13. Secondary Outcome: Relationship to Vaccine of Any Non-serious AEs
Description: Presentation of non-serious AEs by relationship to study vaccine
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Number; unit: Events
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 220 | 208 | 196 | 213
Events
  Unrelated/None | 94 | 67 | 110 | 102
  Unlikely | 24 | 19 | 29 | 23
  Possible | 27 | 15 | 18 | 30
  Probable | 5 | 1 | 0 | 6
  Definite | 107 | 56 | 9 | 34

14. Secondary Outcome: Intensity of Any Non-serious AEs
Description: Presentation of non-serious AEs by intensity
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Number; unit: Events
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 220 | 208 | 196 | 213
Events
  Mild | 233 | 141 | 143 | 163
  Moderate | 20 | 16 | 18 | 25
  Severe | 4 | 1 | 5 | 7

15. Secondary Outcome: Solicited General AEs
Description: Occurrence, intensity and relationship of solicited general AEs (body temperature [fever], headache, myalgia [muscle pain], chills, nausea, fatigue, malaise)
Time Frame: within 15 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 208 | 193 | 187 | 200
Participants
  Pyrexia, Grade 1, Related | 0 | 0 | 0 | 1
  Pyrexia, Grade 2, Related | 2 | 0 | 1 | 1
  Pyrexia, Grade 3, Related | 0 | 1 | 0 | 1
  Headache, Grade 1, Related | 25 | 11 | 17 | 38
  Headache, Grade 2, Related | 6 | 3 | 7 | 21
  Headache, Grade 3, Related | 1 | 2 | 1 | 9
  Myalgia, Grade 1, Related | 28 | 13 | 15 | 44
  Myalgia, Grade 2, Related | 5 | 5 | 2 | 21
  Myalgia, Grade 3, Related | 0 | 1 | 0 | 7
  Chills, Grade 1, Related | 1 | 0 | 8 | 19
  Chills, Grade 2, Related | 0 | 2 | 2 | 12
  Chills, Grade 3, Related | 1 | 0 | 0 | 2
  Nausea, Grade 1, Related | 7 | 4 | 6 | 21
  Nausea, Grade 2, Related | 0 | 2 | 4 | 12
  Nausea, Grade 3, Related | 1 | 0 | 1 | 6
  Fatigue, Grade 1, Related | 29 | 14 | 21 | 45
  Fatigue, Grade 2, Related | 7 | 2 | 7 | 30
  Fatigue, Grade 3, Related | 1 | 1 | 1 | 8
  Malaise, Grade 1, Related | 16 | 6 | 12 | 30
  Malaise, Grade 2, Related | 5 | 2 | 8 | 25
  Malaise, Grade 3, Related | 2 | 1 | 2 | 10

16. Secondary Outcome: Incidence of Lymphadenopathy
Description: Incidence of events of Lymphadenopathy. Pooled solicited and unsolicited events.
Time Frame: within 29 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 220 | 208 | 196 | 213
Participants | 24 | 15 | 17 | 109

17. Secondary Outcome: Solicited Local AEs: Intensity
Description: Incidence of solicited local AEs (pain, redness [erythema], swelling, induration, itching [pruritus])
Time Frame: within 15 days after vaccination
Population: Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
Number analyzed (Participants) | 208 | 193 | 187 | 200
Participants
  Injection Site Pain, Grade 1 | 72 | 49 | 21 | 58
  Injection Site Pain, Grade 2 | 21 | 22 | 6 | 44
  Injection Site Pain, Grade 3 | 4 | 0 | 1 | 33
  Injection Site Erythema, Grade 1 | 44 | 40 | 106 | 105
  Injection Site Erythema, Grade 2 | 9 | 10 | 9 | 81
  Injection Site Erythema, Grade 3 | 0 | 0 | 0 | 5
  Injection Site Swelling, Grade 1 | 14 | 16 | 46 | 120
  Injection Site Swelling, Grade 2 | 5 | 6 | 0 | 17
  Injection Site Swelling, Grade 3 | 0 | 0 | 0 | 1
  Injection Site Induration, Grade 1 | 23 | 11 | 44 | 125
  Injection Site Induration, Grade 2 | 1 | 2 | 1 | 7
  Injection Site Induration, Grade 3 | 0 | 0 | 0 | 0
  Injection Site Pruritus, Grade 1 | 24 | 19 | 99 | 101
  Injection Site Pruritus, Grade 2 | 3 | 1 | 11 | 60
  Injection Site Pruritus, Grade 3 | 2 | 0 | 1 | 18

18. Secondary Outcome: Major Lesion Size, Major Erythema, and Major Induration Diameter
Description: Daily measurement of major lesion size, major erythema, and major induration diameter (mm) based on physical appearance of vaccination site as documented in the memory aid. If the shape of the lesion, erythema [excludes lymphangitis], and induration observed was not round but rather asymmetrical, then the largest [or major] cross-sectional measurement was recorded.
Time Frame: Within 15 days after scarification with ACAM2000
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: mm
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 220 | 213
mm
  Maximum Lesion Diameter | 5.0 [4.0 to 5.0] | 11.5 [11.0 to 12.0]
  Maximum Erythema | 6.0 [5.0 to 7.0] | 26.0 [25.0 to 30.0]
  Maximum Induration | 5.0 [4.0 to 9.0] | 15.0 [13.0 to 16.0]

19. Secondary Outcome: GMTs at the Peak Visits and Individual Peak Measured by Vaccinia-specific ELISA
Description: Peak Visit was defined as Day 42 for Group 1 and Day 28 for Group 2. Individual Peak was the maximum titer per subject from Visit 1 to Visit 7 (Week 8) in Group 1 and maximum titer from Visit 1 to Visit 6 (Week 8) in Group 2.
  Titers below the detection limit are included with a value of 1.
Time Frame: within 8 weeks (for both groups)
Population: Per-protocol Set for Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
Titer
  Peak Visit | 1076.9 [956.8 to 1212.0] | 194.6 [162.6 to 232.9]
  Individual Peak | 1105.2 [983.4 to 1242.0] | 214.0 [177.8 to 257.6]

20. Secondary Outcome: GMTs at the Individual Peak Measured by Vaccinia-specific PRNT
Description: Individual Peak was the maximum titer per subject from Visit 1 to Visit 7 (Week 8) in Group 1 and maximum titer from Visit 1 to Visit 6 (Week 8) in Group 2.
  Titers below the detection limit are included with a value of 1.
Time Frame: within 8 weeks (for both groups)
Population: Per-protocol Set for Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
Titer | 201.5 [178.5 to 227.5] | 117.8 [102.3 to 135.7]

21. Secondary Outcome: GMTs as Measured by Vaccinia-specific ELISA
Description: GMT based on vaccinia-specific ELISA. Titers below the detection limit are included with a value of '1'.
Time Frame: within 12 weeks
Population: Per-protocol Set for Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
Titer
  Week 0 | 1.2 [1.1 to 1.3] | 1.2 [1.0 to 1.3]
  Week 1 | 1.6 [1.3 to 2.0] | 1.2 [1.0 to 1.3]
  Week 2 | 104.9 [84.0 to 131.0] | 21.9 [15.9 to 30.2]
  Week 4 | 129.8 [107.1 to 157.2] | 194.6 [162.6 to 232.9]
  Week 6 | 1076.9 [956.8 to 1212.0] | 149.2 [123.6 to 180.1]
  Week 8 | 671.9 [597.2 to 755.8] | 113.7 [93.2 to 138.7]
  Week 12 | 550.5 [482.2 to 628.4] | NA [NA to NA] — No week 12 visit for Group 2

22. Secondary Outcome: GMTs as Measured by Vaccinia-specific PRNT
Description: GMT based on vaccinia-specific PRNT. Titers below the detection limit are included with a value of '1'.
Time Frame: within 12 weeks
Population: Per-protocol Set for Immunogenicity
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
Titer
  Week 0 | 1.0 [1.0 to 1.1] | 1.0 [1.0 to 1.0]
  Week 1 | 1.1 [1.0 to 1.3] | 1.0 [1.0 to 1.0]
  Week 2 | 16.2 [13.0 to 20.1] | 16.2 [13.1 to 20.0]
  Week 4 | 16.9 [13.7 to 20.8] | 79.3 [67.1 to 93.8]
  Week 6 | 153.5 [134.3 to 175.6] | 64.7 [54.9 to 76.2]
  Week 8 | 118.2 [102.9 to 135.8] | 67.1 [56.9 to 79.0]
  Week 12 | 96.5 [80.1 to 116.2] | NA [NA to NA] — No week 12 visit for Group 2

23. Secondary Outcome: PRNT Seroconversion Rates at Peak Visits
Description: Seroconversion rate based on PRNT. Seroconversion is defined as the appearance of antibody titers "greater than or equal" detection limit (2) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: Group 1 at Week 6; Group 2 at Week 4
Population: Per-protocol Set for Immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
percentage of subjects | 100.0 [98.0 to 100.0] | 97.3 [93.8 to 99.1]

24. Secondary Outcome: ELISA Seroconversion Rates at Peak Visits
Description: Seroconversion rate based on ELISA. Seroconversion is defined as the appearance of antibody titers "greater than or equal" detection limit (50) for initially seronegative subjects, or a doubling or more of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: Group 1 at Week 6; Group 2 at Week 4
Population: Per-protocol Set for Immunogenicity
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 185 | 186
percentage of subjects | 100 [98.0 to 100.0] | 96.8 [93.1 to 98.8]

ADVERSE EVENTS:
Time Frame: 38 weeks for Group 1 and 30 weeks for Group 2
Arm/Group | Group 1, Period 1 | Group 1, Period 2 | Group 1, Period 3 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/208 | 0/196 | 0/213
Serious Adverse Events (participants affected / at risk) | 2/220 | 0/208 | 3/196 | 3/213
Other Adverse Events (participants affected / at risk) | 95/220 | 63/208 | 79/196 | 88/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1, Period 1 (N=220) | Group 1, Period 2 (N=208) | Group 1, Period 3 (N=196) | Group 2 (N=213)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonsillar Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1, Period 1 (N=220) | Group 1, Period 2 (N=208) | Group 1, Period 3 (N=196) | Group 2 (N=213)
Lymphadenopathy (Blood and lymphatic system disorders) | 10 (11) | 6 (6) | 3 (3) | 23 (27)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Injection Site Erythema (General disorders) | 30 (30) | 23 (23) | 1 (1) | 0 (0)
Injection Site Nodule (General disorders) | 32 (38) | 13 (13) | 1 (1) | 0 (0)
Vaccination Site Erythema (General disorders) | 10 (10) | 7 (7) | 2 (2) | 0 (0)
Vaccination Site Nodule (General disorders) | 11 (11) | 3 (3) | 0 (0) | 2 (2)
Vaccination Site Warmth (General disorders) | 13 (13) | 10 (10) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 7 (7) | 4 (4) | 6 (6) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 14 (14) | 14 (14) | 14 (14) | 14 (14)
Laceration (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 2 (2) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 6 (6) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 44 (44) | 49 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Statistical Analysis Plan: Edition 8 (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT01913353/SAP_000.pdf
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT01913353/Prot_001.pdf
  • Statistical Analysis Plan: Edition 8, Amendment 1 (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT01913353/SAP_002.pdf